CLINICAL TRIAL: NCT06869720
Title: The Impact of Eecentric Exercise on Cardiopulmonary Fitness and Quality of Life in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Eecentric Exercise on Cardiopulmonary Fitness and Quality of Life With Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to persistent challenges in participant recruitment, the study has been terminated and the protocol has been formally withdrawn.
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Assistant Professor, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FJUH113384
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-03

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Pulmonary rehabilitation; Eccentric exercise; Chronic obstructive pulmonary disease; Cardiopulmonary fitness; Functional fitness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: eccentric cycling exercise (Experimental): Received eccentric cycling exercise
  Interventions: Device: Eccentric bike
- Control group (Active Comparator): Undergoing conventional treatment
  Interventions: Other: conventional group

INTERVENTIONS:
Device: Eccentric bike — Received eccentric cycling exercise
  Arms: Intervention Group: eccentric cycling exercise
Other: conventional group — Received conventional treatment
  Arms: Control group

SUMMARY:
This study aims to investigate the effects of elliptical exercise on the six-minute walk test and quality of life in patients with chronic obstructive pulmonary disease (COPD) to identify the most efficient exercise training method.

DETAILED DESCRIPTION:
Background： Chronic respiratory diseases, including COPD, are leading causes of chronic illness and mortality worldwide. However, limitations in ventilation and muscle function restrict COPD patients from engaging in higher-power exercise therapies. Compared to concentric exercise, eccentric exercise can effectively improve health-related fitness and quality of life at lower cardiopulmonary and metabolic loads. Pulmonary rehabilitation programs have been shown to effectively improve symptoms of chronic respiratory diseases, increase exercise capacity, enhance quality of life, delay disease progression, prevent and treat acute exacerbations, and reduce mortality. Therefore, it is hoped that a "safe and effective" eccentric exercise strategy can be designed for COPD patients to comprehensively improve their cardiopulmonary/muscle fitness and quality of life, thereby improving the course of their disease.

Study Design： This is a one-year, single-center, prospective randomized controlled trial. Methods： This study plans to enroll 60 participants who will be randomly assigned to control and experimental groups. The intervention will take place in the pulmonary rehabilitation room on the sixth floor of Fu Jen Hospital. Each group will undergo a functional fitness test and complete a quality of life questionnaire before and after 24 sessions (over 12 weeks) of exercise training.

Effect： It is anticipated that after 24 sessions of elliptical exercise training, there will be an improvement in the functional fitness and in quality of life related to physical activity function.

Key words： Pulmonary rehabilitation; eccentric exercise; chronic obstructive pulmonary disease; cardiopulmonary fitness; functional fitness

ELIGIBILITY:
Inclusion Criteria:

* Having undergone pulmonary rehabilitation for more than 3 months
* Sign the written informed consent form
* FEV1/FVC < 0.70
* Approval for exercise training granted by a specialist physician's assessment
* Specialist physician's approval for exercise training

Exclusion Criteria:

* Existing of tracheostomy
* Those who use oxygen therapy or ventilator at home
* Severe heart failure (NYHA III-IV)
* Neuromuscular disease
* Acute exacerbation within the past three months
* Those who are unable to cooperate with the cardiopulmonary exercise test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
six minute walk test | 12 weeks
  functional performance
time up and go | 12 weeks
  functional performance
stairs ascending and descending walking time | 12 weeks
  functional performance

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No